CLINICAL TRIAL: NCT02688231
Title: Intensity Dependent Clinical Effects of a Task-oriented Upper Limb Training in Multiple Sclerosis
Brief Title: Task-oriented Upper Limb Training in MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Peter Feys, Professor, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S58587
Record Dates: First submitted 2016-02-09; First posted 2016-02-23 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Upper limb rehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High intensity group (Experimental)
  Interventions: Other: Task-oriented upper limb training
- Low intensity group (Experimental)
  Interventions: Other: Task-oriented upper limb training
- Control group - conventional treatment (Active Comparator)
  Interventions: Other: Control intervention

INTERVENTIONS:
Other: Task-oriented upper limb training — Participants in the experimental groups (high-intensity and low-intensity) receive for 8 weeks, 60 min/day, 5 days/week a task-oriented upper limb rehabilitation training at a high or low intensity, respectively, instead of their regular occupational therapy hours provided in the conventional multidisciplinary rehabilitation program.
  The task-oriented training involves practicing of functional daily tasks, with the intention to acquire or reacquire a skill. Most functional upper limb tasks require following essential movement components: reaching, moving, positioning, transporting, lifting the upper limb and/or an object and grasping, releasing, stabilizing, manipulating an object.
  The Tagtrainer of SymbioTherapy is used to support the independent training of tasks with real objects with different sizes and weights. The Diego of Tyromotion is used in patients who require assistance (gravity support) during the performance of different upper limb tasks.
  Arms: High intensity group; Low intensity group
Other: Control intervention — The participants in the control group receive for 8 weeks the conventional multidisciplinary rehabilitation program (physiotherapy, occupational therapy and speech or cognitive therapy if needed).
  The training sessions are scheduled for 60 min/day, 5 days/week for the duration of 8 weeks.
  Arms: Control group - conventional treatment

SUMMARY:
An adequate upper limb function is crucial to independently perform Activities of Daily Living (ADL). Persons with neurological diseases often experience upper limb dysfunction. Upper limb function in Multiple Sclerosis (MS) is highly prevalent, increasing with overall disability level, while the detrimental impact on ADL is higher than in stroke, given that symptoms often occur bilaterally. In contrast to stroke, it is unknown whether similar rehabilitation principles and effect sizes apply in MS given that this progressive neurodegenerative disease is characterized by multiple lesions and atrophy of brain structures. To date, optimal therapy dosage of upper limb rehabilitation programs are not known in the MS literature neither were characteristics of responders identified.

The aim of this explorative study is to investigate the intensity dependent clinical effects of a task-oriented upper limb training in persons with MS with different upper limb disability levels.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of MS (McDonald criteria)
* Progressive type of MS (primary or secondary progressive MS)
* A score 1 or more on the performance scale: item hand function

Exclusion Criteria:

* A relapse or relapse-related treatment within the last 3 months prior to the study
* Complete paralysis of both upper limbs
* Marked or severe intention tremor (Fahn's tremor rating scale > 3)
* Other medical conditions interfering with the upper limb function (ortopaedic or rheumatoid impairment)
* Severe cognitive or visual deficits interfering with testing and training

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Nine Hole peg test | 8 weeks
  Manual dexterity
Manual Ability Measure-36 | 8 weeks
  Questionnaire about perceived ADL performance
Isometric hand grip | 8 weeks
  Isometric hand grip
Training tolerance | daily through study compeletion
  Questionnaire of training tolerance and possible adverse effects
pinch grip strength | 8 weeks
  pinch grip strength

SECONDARY OUTCOMES:
Motricity Index | 8 weeks
  General isometric muscle strength
Muscle fatigue indices | 8 weeks
  Indices calculated based on a 30 seconds sustained maximal isometric hand grip contraction
Tactile sensitivity in the fingers Semmens-Weinstein monofilaments | 8 weeks
  Tactile sensitivity in the thumb and index
Rydel Seiffer Tuning fork | 8 weeks
  Vibration in the upper limb
Symbol digit modalities test | 8 weeks
  Cognitive function, processing speed
Box and block test | 8 weeks
  Manual dexterity
Action Research Arm Test | 8 weeks
  Proximal and distal upper limb function
Test d'Évaluation des Membres Supérieurs des Personnes Âgées (TEMPA) | 8 weeks
  Proximal and distal upper limb function
Virtual Peg Insertion Test | 8 weeks
  manual dexterity
Accelerometers (Actigraph) | 8 weeks
  actual upper limb performance in daily life

CONTACTS AND LOCATIONS:
Overall Officials: Peter Feys, Prof. dr., Principal Investigator — REVAL - Rehabilitation Research Center, BIOMED - Biomedical Research Institute, Faculty of Medicine and Life Sciences, Hasselt University, Hasselt, Belgium
Locations (2):
- Belgium (2):
  - Revalidatie en MS centrum, Overpelt, Limburg
  - Hasselt University, Diepenbeek

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lamers I, Maris A, Severijns D, Dielkens W, Geurts S, Van Wijmeersch B, Feys P. Upper Limb Rehabilitation in People With Multiple Sclerosis: A Systematic Review. Neurorehabil Neural Repair. 2016 Sep;30(8):773-93. doi: 10.1177/1545968315624785. Epub 2016 Jan 7. PMID 26747125
- [Background] Severijns D, Octavia JR, Kerkhofs L, Coninx K, Lamers I, Feys P. Investigation of Fatigability during Repetitive Robot-Mediated Arm Training in People with Multiple Sclerosis. PLoS One. 2015 Jul 27;10(7):e0133729. doi: 10.1371/journal.pone.0133729. eCollection 2015. PMID 26213990
- [Background] Feys P, Coninx K, Kerkhofs L, De Weyer T, Truyens V, Maris A, Lamers I. Robot-supported upper limb training in a virtual learning environment : a pilot randomized controlled trial in persons with MS. J Neuroeng Rehabil. 2015 Jul 23;12:60. doi: 10.1186/s12984-015-0043-3. PMID 26202325
- [Background] Alt Murphy M, Resteghini C, Feys P, Lamers I. An overview of systematic reviews on upper extremity outcome measures after stroke. BMC Neurol. 2015 Mar 11;15:29. doi: 10.1186/s12883-015-0292-6. PMID 25880033
- [Background] Bertoni R, Lamers I, Chen CC, Feys P, Cattaneo D. Unilateral and bilateral upper limb dysfunction at body functions, activity and participation levels in people with multiple sclerosis. Mult Scler. 2015 Oct;21(12):1566-74. doi: 10.1177/1352458514567553. Epub 2015 Feb 6. PMID 25662346
- [Background] Severijns D, Lamers I, Kerkhofs L, Feys P. Hand grip fatigability in persons with multiple sclerosis according to hand dominance and disease progression. J Rehabil Med. 2015 Feb;47(2):154-60. doi: 10.2340/16501977-1897. PMID 25268997
- [Background] Lamers I, Cattaneo D, Chen CC, Bertoni R, Van Wijmeersch B, Feys P. Associations of upper limb disability measures on different levels of the International Classification of Functioning, Disability and Health in people with multiple sclerosis. Phys Ther. 2015 Jan;95(1):65-75. doi: 10.2522/ptj.20130588. Epub 2014 Sep 4. PMID 25190063
- [Background] Lamers I, Feys P. Assessing upper limb function in multiple sclerosis. Mult Scler. 2014 Jun;20(7):775-84. doi: 10.1177/1352458514525677. Epub 2014 Mar 24. PMID 24664300
- [Background] Lamers I, Kelchtermans S, Baert I, Feys P. Upper limb assessment in multiple sclerosis: a systematic review of outcome measures and their psychometric properties. Arch Phys Med Rehabil. 2014 Jun;95(6):1184-200. doi: 10.1016/j.apmr.2014.02.023. Epub 2014 Mar 13. PMID 24631802
- [Background] Lambercy O, Fluet MC, Lamers I, Kerkhofs L, Feys P, Gassert R. Assessment of upper limb motor function in patients with multiple sclerosis using the Virtual Peg Insertion Test: a pilot study. IEEE Int Conf Rehabil Robot. 2013 Jun;2013:6650494. doi: 10.1109/ICORR.2013.6650494. PMID 24187309
- [Background] Lamers I, Timmermans AA, Kerkhofs L, Severijns D, Van Wijmeersch B, Feys P. Self-reported use of the upper limbs related to clinical tests in persons with multiple sclerosis. Disabil Rehabil. 2013;35(23):2016-20. doi: 10.3109/09638288.2013.771703. Epub 2013 Apr 29. PMID 23627537
- [Background] Lamers I, Kerkhofs L, Raats J, Kos D, Van Wijmeersch B, Feys P. Perceived and actual arm performance in multiple sclerosis: relationship with clinical tests according to hand dominance. Mult Scler. 2013 Sep;19(10):1341-8. doi: 10.1177/1352458513475832. Epub 2013 Feb 13. PMID 23407701
- [Background] van den Hoogen W, Feys P, Lamers I, Coninx K, Notelaers S, Kerkhofs L, Ijsselsteijn W. Visualizing the third dimension in virtual training environments for neurologically impaired persons: beneficial or disruptive? J Neuroeng Rehabil. 2012 Oct 5;9:73. doi: 10.1186/1743-0003-9-73. PMID 23036010
- [Background] Broekmans T, Gijbels D, Eijnde BO, Alders G, Lamers I, Roelants M, Feys P. The relationship between upper leg muscle strength and walking capacity in persons with multiple sclerosis. Mult Scler. 2013 Jan;19(1):112-9. doi: 10.1177/1352458512444497. Epub 2012 May 4. PMID 22562952
- [Background] Gijbels D, Lamers I, Kerkhofs L, Alders G, Knippenberg E, Feys P. The Armeo Spring as training tool to improve upper limb functionality in multiple sclerosis: a pilot study. J Neuroeng Rehabil. 2011 Jan 24;8:5. doi: 10.1186/1743-0003-8-5. PMID 21261965
- [Derived] Lamers I, Raats J, Spaas J, Meuleman M, Kerkhofs L, Schouteden S, Feys P. Intensity-dependent clinical effects of an individualized technology-supported task-oriented upper limb training program in Multiple Sclerosis: A pilot randomized controlled trial. Mult Scler Relat Disord. 2019 Sep;34:119-127. doi: 10.1016/j.msard.2019.06.014. Epub 2019 Jun 17. PMID 31255988